CLINICAL TRIAL: NCT05494671
Title: Studying Corneal Epithelial Stability Following Limbal Stem Cell Transplantation in Cases of Limbal Stem Cell Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fayrouz Aboalazayem, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N-14-2022
Record Dates: First submitted 2022-08-07; First posted 2022-08-10 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Stem Cell Transplantation
Keywords: stem cell transplantation,; stem cell deficiency; CLAU

STUDY DESIGN:
Intervention Model Description: interventional case series
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- conjunctival limbal autologous transplant (Experimental): patients with unilateral stem cell deficiency due to chemical burn
  Interventions: Procedure: conjunctival limbal autologous transplant

INTERVENTIONS:
Procedure: conjunctival limbal autologous transplant — Patients with unilateral chemical ocular injury will be included in the study. All selected patients will receive a thorough explanation of the study design and aims and informed consent will be obtained in all patients. Eyes of all participants will be subjected to: Best corrected visual acuity, Slit lamp examination and ocular ultrasound if no fundus view.
  Staging of degree of limbal stem cell deficiency is done by Roper Hall classification and then the patient will have conjunctival limbal autologous transplant (CLAU)

SUMMARY:
Integrity of the corneal epithelium is the function of intact limbal stem cells. The reduction in the population of LSCs and their dysfunction result in abnormal corneal epithelialization and invasion of the corneal surface by the conjunctival epithelium with or without corneal neovascularization that is, limbal stem cell deficiency (LSCD). Different techniques have been developed to treat cases of limbal stem cell deficiency due to traumatic or congenital cases. Recent innovations developed to predict the early stages of stem cell deficiency. One of these methods is measurement of the central epithelial thickness as it was found that limbal stem cell deficiency causes reduction of the central epithelial thickness.

The aim of this study is to study changes in the corneal epithelial thickness at different quadrants of the cornea to observe the exact time of epithelial stability following stem cell transplantation.

DETAILED DESCRIPTION:
Patients with unilateral chemical ocular injury will be included in the study(12 eyes). All selected patients will receive a thorough explanation of the study design and aims and informed consent will be obtained in all patients. Eyes of all participants will be subjected to: Best corrected visual acuity, Slit lamp examination and ocular ultrasound if no fundus view.

Staging of degree of limbal stem cell deficiency is done by Roper Hall classification and then the patient will have conjunctival limbal autologous transplant (CLAU).

The patient will be followed up at a week, a month, 3 months, 6months and 9 months postoperative.

Corneal epithelial mapping will be done at the previous schedule in both the donated and the recipient eyes using anterior segment OCT (Optical Coherence Tomography)

Exclusion criteria:

Bilateral cases and patients with severe conjunctival scaring and symblepharon.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 15 to 70 years
* Unilateral limbal stem cell deficiency
* Grade 4 stem cell deficiency

Exclusion Criteria:

* Cases with extensive symblepharon
* Cases with very poor visual acuity ( no light perception)
* Cases with posterior segment problem evident in ocular ultrasonography

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
the change of corneal epithelial thickness after stem cell transplantation over 9 months | 9 months
  Corneal epithelial mapping will be done at one month, 3,6 and 9 months in both the donated and the recipient eyes using anterior segment OCT at the center

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Egypt